CLINICAL TRIAL: NCT03374449
Title: Impact of Renin-Angiotensin System Inhibitors Continuation on Outcome After Major Surgery : a Multicenter, Prospective, Randomized and Controlled Trial
Brief Title: Impact of Renin-Angiotensin System Inhibitors Continuation on Outcome After Major Surgery
Acronym: STOPORNOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P160933J
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Renin Angiotensin System; Surgery
Keywords: Major surgery; Postoperative morbidity and mortality; Renin angiotensin system inhibitors

STUDY DESIGN:
Intervention Model Description: The aim of this study is to evaluate the impact of Renin-Angiotensin System inhibitors management (Continuation or discontinuation 48 hours before surgery) on outcome in patients undergoing scheduled major non-cardiac surgery (surgery with an expected duration of more than 2 hours from the surgical incision and a post-operative hospital stay of least 3 days)
Masking Description: Endpoint validated by an adjudication commitee blinded to the arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuation of the RAS-inhibitors (Experimental): in the continuation of the RAS-inhibitors arm the treatment will be continued until the morning the day of surgery.
  Interventions: Procedure: continuation of the RAS-inhibitors
- discontinuation of the RAS-inhibitors (Active Comparator): In this arm : discontinuation of the RAS-inhibitors 48 hours before surgery Patients won't receive the drug on the morning of the day of the surgery.
  Interventions: Procedure: discontinuation of the RAS-inhibitors

INTERVENTIONS:
Procedure: continuation of the RAS-inhibitors — drug intake
  Arms: continuation of the RAS-inhibitors
Procedure: discontinuation of the RAS-inhibitors — no drug intake
  Arms: discontinuation of the RAS-inhibitors

SUMMARY:
More than 200 million major surgical procedures are performed annually worldwide. Many of these patients have comorbidities including hypertension and/or heart failure. Chronic treatment of hypertension and/or heart failure very often includes a Renin-Angiotensin System (RAS) inhibitor (Angiotensin-Converting Enzyme Inhibitors (ACE-Is) or Angiotensin Receptor Blockers (ARBs). To stop or not to stop these medications before major surgery remain unknown. Data on management of RAS inhibitors before major surgery and anesthesia remain lacking and matter of debate. It is much likely that the strategy regarding management of RAS inhibitors in the peri-operative setting have important impact on peri-operative complications.

The lack of evidence leads to conflicting guidelines with respect to RAS inhibitors management before major surgery. While French guidelines are to stop RAS inhibitors patients with hypertension to avoid profound anesthestic-drugs-induced hypotension, international guidelines differ. The American heart association task force states that continuation of RAS inhibitors perioperatively is reasonable (class IIa recommendation,level of evidence: B). The purpose of this study is to determine the prognostic impact of withholding vs continuing ARBs before major non cardiac surgery.

DETAILED DESCRIPTION:
Multicenter, prospective, randomized, pragmatic, parallel-group clinical trial. The inclusion visit takes place between 4 months and no later than 3 days before the surgery visit.

* The randomization will be performed by the anesthesiologist Control group : RAS-I discontinuation Experimental group: RAS-I continuation
* A prescription for the medication strategy (stopping or pursuing the medication) will be handed to the patient during the anesthesiology consultation.

Five follow-up visits are planned

* Immediately, one hour after the surgery (Day 0)
* Then four follow-up visits are planned on day 1, 2, 7 (or hospital discharge) and 28 days+15 days (43 days maximum) after surgery will be collected data and parameters for study endpoints.

End of research visit is the 28 days+15 days (43 days maximum) follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring major non-cardiac surgery (surgery with an expected duration of more than 2 hours from the surgical incision and a post-operative hospital stay of least 3 days) (according to the study RELIEF, DOI : 10.1056/NEJMoa1801601))
* Age≥18 years
* Patients chronically treated (>3 months before surgery) with RAS inhibitors
* Pregnancy test at inclusion visit for women of childbearing potential Women of childbearing potential must agree to use adequate contraception according to Recommendations related to contraception and pregnancy testing in clinical trials, by Clinical Trial Facilitation Group (CTFG)
* Signed informed consent

Exclusion Criteria:

* Emergency surgery (surgical treatment needed within 24 hours)
* Hyperkalemia (> 5.5mmol/L) known at the time of the anesthetic consultation
* Patients for which death is deemed imminent and inevitable or patients with an underlying disease process with a life expectancy of less than 1 month
* Patient with severe renal insufficiency, known at the time of the anesthestic consultation (as defined by estimated glomerular filtration rate (creatinine clearance <15 ml/min/1.73m2 or requiring renal replacement therapy)
* Patient with preoperative shock (defined by the need for vasoactive drugs before surgery)
* Inability to obtain informed consent either from the patient.
* Lack of Social Insurance

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2222 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
composite outcome composed of all-cause mortality and major postoperative complications within 28 days after surgery. | after surgery until day 28
  Complications will be validated by an adjudication committee, blinded to the treatment arm.
  Death; Acute Myocardial infarction; Arterial or venous thrombosis; Stroke; Acute pulmonary oedema; Post-operative cardiogenic shock; Acute severe hypertension crisis; Cardiac arrhythmia requiring therapeutic intervention; Postoperative episodes of sepsis; Postoperative respiratory complication; Need for unplanned intensive care unit admission or readmission; Acute kidney injury: KDIGO criteria Baseline serum creatinine is obtained from the pre-operative blood sample; Surgical complications: need for reoperation for any reason and radiologic interventions for abscess drainage; Severe Hyperkalemia: serum potassium level >5.5 mmol/L and requiring therapeutic intervention (insulin/glucose infusion and/or sodium bicarbonate infusion and/or intravenous B2 agonists and/or intravenous calcium gluconate and/or renal replacement therapy and/or ventricular tachycardia or ventricular fibrillation).

SECONDARY OUTCOMES:
Episodes of hypotension | during anesthesia and surgery
  Episodes requiring vasopressors administration
Acute kidney injury | after surgery until day 28
  according to the KDIGO criteria
Maximum SOFA score | from postoperative day 1 to day 7
  patients admitted to ICU
Duration of hospital stay | after surgery until day 28
  Patients who will be outside the hospital but in other types of health care facilities at day 28 will be considered to have been discharged home
Hospital free-days | censored at 28 days following surgery
  Duration after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Eienne Gayat, MD, PhD, Principal Investigator — Hospital Laribioisière, APHP
Locations (1):
- Hospital Lariboisiere, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legrand M, Payen D. Case scenario: Hemodynamic management of postoperative acute kidney injury. Anesthesiology. 2013 Jun;118(6):1446-54. doi: 10.1097/ALN.0b013e3182923e8a. No abstract available. PMID 23558177
- [Background] Augoustides JG. Angiotensin blockade and general anesthesia: so little known, so far to go. J Cardiothorac Vasc Anesth. 2008 Apr;22(2):177-9. doi: 10.1053/j.jvca.2008.01.002. No abstract available. PMID 18375316
- [Background] Mets B. To stop or not? Anesth Analg. 2015 Jun;120(6):1413-9. doi: 10.1213/ANE.0000000000000758. No abstract available. PMID 25988640
- [Background] Mets B, Hennrikus E. Perioperative angiotensin axis blockade, to continue or discontinue, that is the question? Anesth Analg. 2014 Nov;119(5):1223-4. doi: 10.1213/ANE.0000000000000430. No abstract available. PMID 25329033
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN; American College of Cardiology; American Heart Association. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines. J Am Coll Cardiol. 2014 Dec 9;64(22):e77-137. doi: 10.1016/j.jacc.2014.07.944. Epub 2014 Aug 1. No abstract available. PMID 25091544
- [Derived] Pirracchio R, Cholley B, Falcone J, Charbonneau H, Delaporte A, Lemoine A, Joosten A, Gayat E, Legrand M; STOP-or-NOT trial group. Impact of continuing renin-angiotensin-aldosterone system inhibitors before surgery on intraoperative hypotensive events: a secondary analysis of the STOP-or-NOT Trial. Br J Anaesth. 2026 Jan 8:S0007-0912(25)00860-8. doi: 10.1016/j.bja.2025.11.049. Online ahead of print. PMID 41513520
- [Derived] Tang J, Pirracchio R, Cholley B, Joosten A, Birckener J, Falcone J, Charbonneau H, Delaporte A, Chen D, Gayat E, Legrand M. Preoperative Cardiovascular Risk and Postoperative Outcomes by Renin-Angiotensin System Inhibitor Use: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2025 Sep 1;10(9):942-948. doi: 10.1001/jamacardio.2025.1920. PMID 40560582
- [Derived] Legrand M, Falcone J, Cholley B, Charbonneau H, Delaporte A, Lemoine A, Garot M, Joosten A, Meistelman C, Cheron-Leroy D, Rives JP, Pastene B, Dewitte A, Sigaut S, Danguy des Deserts M, Truc C, Boisson M, Lasocki S, Cuvillon P, Schiff U, Jaber S, Le Guen M, Caillard A, Bar S, Pereira de Souza Neto E, Colas V, Dimache F, Girardot T, Jozefowicz E, Viquesnel S, Berthier F, Vicaut E, Gayat E; Stop-or-Not Trial Group. Continuation vs Discontinuation of Renin-Angiotensin System Inhibitors Before Major Noncardiac Surgery: The Stop-or-Not Randomized Clinical Trial. JAMA. 2024 Sep 24;332(12):970-978. doi: 10.1001/jama.2024.17123. PMID 39212270
- [Derived] Legrand M, Futier E, Leone M, Deniau B, Mebazaa A, Plaud B, Coriat P, Rossignol P, Vicaut E, Gayat E; STOP-OR-NOT study investigators. Impact of renin-angiotensin system inhibitors continuation versus discontinuation on outcome after major surgery: protocol of a multicenter randomized, controlled trial (STOP-or-NOT trial). Trials. 2019 Mar 5;20(1):160. doi: 10.1186/s13063-019-3247-1. PMID 30836981